CLINICAL TRIAL: NCT03033290
Title: Effect of Traditional Chinese Medicine on Gut Microbiota, Physical Constitution, and Allergic Diseases
Brief Title: Traditional Chinese Medicine on Gut Microbiota and Allergic Diseases
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, YANG SIEN-HUNG, Director of Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CORPG1F0011
Record Dates: First submitted 2016-05-31; First posted 2017-01-26 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Allergic Rhinitis
Keywords: Qi-tonifying regimen; immune-modulation; gut microbiota
MeSH Terms: conditions — Rhinitis, Allergic | interventions — bu-zhong-yi-qi-tang

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bu-Zhong-Yi-Qi-Tang (BZYQT) (Experimental): capsule of BZYQT, 4gm tid, 12gm a day for 2 months
  Interventions: Drug: Bu-Zhong-Yi-Qi-Tang
- placebo control (Placebo Comparator): similar placebo capsule 4gm tid, 12gm a day for 2 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bu-Zhong-Yi-Qi-Tang — Qi-tonifying regimen of traditional Chinese herbal medicine
  Arms: Bu-Zhong-Yi-Qi-Tang (BZYQT)
Drug: placebo — placebo control
  Arms: placebo control

SUMMARY:
Allergic rhinitis is an importance disease in Taiwan with its high incidence about 20-30% and gradually increased annually. However, symptom relapse still bothered the majority of patients though there were certain advances in western medicine. In addition, side effects of western medicine, such as lethargy, mouth dryness were noted. Traditional Chinese medicine, especially qi-tonifying regimen has been used and proved benefit to the allergic diseases by many researchers.This study will provide the evidences of gut microbiota changes and immune-modulatory effects of BZYQT for the treatment of allergic rhinitis.

DETAILED DESCRIPTION:
Recently studies reported that gut microbiota is related to the human immunity modulation of allergic diseases. Investigators are interested to know weather qi-tonifying herbal medicine is through the changes of gut microbiota to modulate human immunity. In this study, a double-blinded, randomized, placebo control design is applied and total 60 perennial allergic rhinitis patients will be enrolled in our study. All subjects will be divided into Bu-Zhong-Yi-Qi-Tang (BZYQT) and placebo control groups, 40 and 20 subjects each. Subjects of BZYQT group will receive capsule of BZYQT, 4gm tid, 12gm a day, while control group will receive similar placebo capsule with same scheme. Total 2 months treatment course will be done. Gut microbiota will be assayed before and after 2 months treatment. Additionally, various parameters for immunologic response will be checked before and after the treatment, including the total IgE amount, the ratio of CD4/CD8 of T lymphocytes, the profile of cytokine such as IL-10 and IL-12 as well as functional change of dendritic cells and T cells. Results will be analyzed statistically including gender analysis. This study will provide the evidences of gut microbiota changes and immune-modulatory effects of BZYQT for the treatment of allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

1. With at least one of the following clinical symptoms: itchy nose, sneeze, rhinorrhea, nasal congestion
2. Diagnosed as intermittent allergic rhinitis (Less than 4 days per week and for less than 4 weeks)
3. CAP panel :allergy to mite
4. Will to complete questionnaires and take medicine as schedule in this study
5. Volunteer for study enrollment and sign inform consent

Exclusion Criteria:

1. Under treatment of western medicine including steroid, antihistamine, leukotriene inhibitor, immunosuppressant or stop above medication less than one month
2. Under acute inflammatory disease such as pneumonia, sinusitis, bronchitis and so on
3. vasomotor type allergic rhinitis
4. history of allergy or adverse effect to Chinese herbs, poor compliance of herbal medicine
5. severe organ function impairment, such as heart failure, liver failure, renal failure (eGFR <60 mL/min/1.73 m2)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes in allergic rhinitis symptom severity | Assessment of symptom severity on Day 0 and 2 months after completing treatment
  Sino-nasal Outcome Test (SNOT-22)

SECONDARY OUTCOMES:
Improvement of fatigue | Assessment of fatigue severity on Day 0 and 2 months after completing treatment
  Fatigue Severity Scale
Improvement of life quality | Assessment of life quality on Day 0 and 2 months after completing treatment
  SF-36
Detection of gut microbiota | Assessment of gut microbiota on Day 0 and 2 months after completing treatment
  use cecal stool DNA purification and quantification of cecal microbiota by quantitative PCR (qPCR). Using V3-V5 16S rRNA amplification; Processing of NGS data; Operational Taxonomic Units (OTUs) cluster; Taxonomic profiling
Change in serum total and mite specific IgE | Assessment of serologic markers on Day 0 and 2 months after completing treatment
  check serum total IgE and mite specific IgE (KIU/l)
T Cells measurement | Assessment of CD4/CD8 on Day 0 and 2 months after completing treatment
  check CD4 / CD8 by flowcytometry
Measurement of cytokines produced by polymorphonuclear leukocytes | Assessment of serologic markers on Day 0 and 2 months after completing treatment
  check sICAM-1,IL-8,PGE2, LTC4
Measurement of cytokines produced by monocytes and lymphocytes | Assessment of serologic markers on Day 0 and 2 months after completing treatment
  IL-4、IL-5、IL-10、IL-13、IFN-γ
Detection of dendritic cell function | Assessment of serologic markers on Day 0 and 2 months after completing treatment
  check IL-10 and IL-12 level

CONTACTS AND LOCATIONS:
Overall Officials: Sien-hung Yang, Ph.D., Study Director — Chang Gung Memorial Hospital, Taoyuan, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hwang BF, Jaakkola JJ, Lee YL, Lin YC, Guo YL. Relation between air pollution and allergic rhinitis in Taiwanese schoolchildren. Respir Res. 2006 Feb 9;7(1):23. doi: 10.1186/1465-9921-7-23. PMID 16469096
- [Background] Yang SH, Hong CY, Yu CL. Decreased serum IgE level, decreased IFN-gamma and IL-5 but increased IL-10 production, and suppressed cyclooxygenase 2 mRNA expression in patients with perennial allergic rhinitis after treatment with a new mixed formula of Chinese herbs. Int Immunopharmacol. 2001 Jun;1(6):1173-82. doi: 10.1016/s1567-5769(01)00051-0. PMID 11407311
- [Background] Yang SH, Hong CY, Yu CL. The stimulatory effects of nasal discharge from patients with perennial allergic rhinitis on normal human neutrophils are normalized after treatment with a new mixed formula of Chinese herbs. Int Immunopharmacol. 2002 Nov;2(12):1627-39. doi: 10.1016/s1567-5769(02)00133-9. PMID 12469937
- [Background] Yang SH, Yu CL, Chen YL, Chiao SL, Chen ML. Traditional Chinese medicine, Xin-yi-san, reduces nasal symptoms of patients with perennial allergic rhinitis by its diverse immunomodulatory effects. Int Immunopharmacol. 2010 Aug;10(8):951-8. doi: 10.1016/j.intimp.2010.05.008. Epub 2010 May 28. PMID 20546945
- [Background] Kuroiwa A, Liou S, Yan H, Eshita A, Naitoh S, Nagayama A. Effect of a traditional Japanese herbal medicine, hochu-ekki-to (Bu-Zhong-Yi-Qi Tang), on immunity in elderly persons. Int Immunopharmacol. 2004 Feb;4(2):317-24. doi: 10.1016/j.intimp.2003.12.004. PMID 14996423
- [Background] Yang SH, Kao TI, Chiang BL, Chen HY, Chen KH, Chen JL. Immune-modulatory effects of bu-zhong-yi-qi-tang in ovalbumin-induced murine model of allergic asthma. PLoS One. 2015 Jun 2;10(6):e0127636. doi: 10.1371/journal.pone.0127636. eCollection 2015. PMID 26035827
- [Result] Xie MQ, Liu J, Long Z, Tian DF, Zhao CQ, Yang PC. Modulation of immune tolerance with a Chinese traditional prescription inhibits allergic rhinitis in mice. N Am J Med Sci. 2011 Nov;3(11):503-7. doi: 10.4297/najms.2011.3503. PMID 22361496